CLINICAL TRIAL: NCT01281800
Title: Cisplatin With Either Alimta or Gemcitabine in Long Infusion for Mesothelioma: A Randomised Phase II Trial (AGILI Trial)
Brief Title: Cisplatin With Alimta or Gemcitabine in Long Infusion for Mesothelioma
Acronym: AGILI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Viljem Kovac, MD, Institute of Oncology Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22k/06/08
Record Dates: First submitted 2011-01-17; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Gemcitabine

ARMS (2):
- Cisplatin with pemetrexed (Active Comparator)
  Interventions: Procedure: Gemcitabine in long infusion
- Cisplatin with gemcitabine in long infusion (Experimental)
  Interventions: Procedure: Gemcitabine in long infusion

INTERVENTIONS:
Procedure: Gemcitabine in long infusion — TREATMENT A:
  Day 1: Pemetrexed 500 mg/m2 Cisplatin 75 mg/m2 Cycle every 3 weeks. Supportive treatment: folic acid [Tifol 400 mg tbl (350-1000 mg), beginning 7 days before CT, every day, till 3 week after the KT], vitamin B-12 [OH-B12 i.m., beginning in 7 days before CT, than at 3. + 6. cycles of KT + 9. week after the KT], corticosteroids, hydration, antiemetic, LMW heparin as thromboprophylaxis.
  In the absence of progression, 4 cycles of chemotherapy with pemetrexed and cisplatin will be given, followed by two additional cycles of pemetrexed as monotherapy.
  TREATMENT B:
  Days 1 and 8: gemcitabine 250 mg/m2 in 6 hours day 2: cisplatin 75 mg/m2 Cycle every 3 weeks. Supportive treatment: corticosteroids, hydration, antiemetics, LMW heparin as thromboprophylaxis.
  In the absence of progression, 4 cycles of chemotherapy with gemcitabine and cisplatin will be given, followed by two additional cycles of gemcitabine alone as monotherapy.

SUMMARY:
This is a randomised Phase II clinical trial to assess and compare efficacy and safety profile of cisplatin and pemetrexed against cisplatin and low-dose gemcitabine in long infusion.

DETAILED DESCRIPTION:
Combination of pemetrexed and cisplatin is now considered the standard systemic treatment for mesothelioma. Three arguments against such a position are: 1. Pemetrexed in combination with cisplatin was registered for mesothelioma on the basis of superiority over cisplatin alone, a clearly suboptimal control arm; 2. Several Phase II trials of gemcitabine in standard doses or as low-dose in long infusion in combination with cisplatin have shown at least comparable activity; 3. Due to high cost, pemetrexed is not available to many patients in countries with limited health care resources. During the past five years, our research team in Ljubljana conducted a Phase II trial of low-dose gemcitabine (250 mg/m2) in 6-hours infusion and cisplatin for patients with mesothelioma. In an unselected population of patients including those in poor performance status, elderly, patients with advanced extrathoracic disease and patients in progression after previous chemotherapy, the response rate was 54%, and median survival was 16.5 months. On the basis of this favourable experience and in search of cost-effective treatment for mesothelioma, we here propose a randomised Phase II clinical trial to compare efficacy and safety profile of cisplatin and pemetrexed against cisplatin and low-dose gemcitabine in long infusion. The primary endpoints are response rate and time to progression; secondary endpoints are survival, toxicity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven mesothelioma. While local histopathology exam is sufficient to register a patient for the trial, all biopsies will be subject to central review (please see Section 5.3.)
* no history of other malignancy; or in complete remission for > 3 years if previously treated for other malignancy;
* chemo-naive;
* performance status ≥ 70% (Karnofsky); or ECOG 0 - 2 ;
* no peripheral neuropathy grade 2 or more (common toxicity criteria - CTC, NCI), unless mechanical in origin;
* no vascular disease grade 2 or more (NCI CTC ver.3);
* hemoglobin > 100 g/L;
* neutrophils > 2.0 g/L;
* platelets > 100 x 109 /L;
* kidney function: creatinine within normal limits + ECC > 60 mL/min; or ECC > 100 mL/min;
* liver function: bilirubin < 1.25 x UNL; AST/ALT < 2 x UNL;
* cardiac compensation;
* no active infection or other serious concomitant disease;
* women are not pregnant
* patient's understanding of the disease and treatment and written informed consent.

Exclusion Criteria:

• significant medical co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | CT measurement of disease will be performed after 2nd cycle of chemotherapy, at the end of the treatment and during follow up period up to progression (total average 8 months)
  Efficacy of the treatment will be measured by response rate (RR) and progression free survival (PFS) using modified RECIST criteria for assessment of response in malignant pleural mesothelioma

SECONDARY OUTCOMES:
Overall survival | Outcome measures will be assessed during average time period of 18 months from enrollment
  Efficacy of the treatment will be measured also by overall survival (OS).
  Safety and tolerability will be assessed by monitoring the adverse events during treatment and follow-up phase and graded according the NCI Common Toxicity Criteria (CTC), version 3.0.
  Quality of life (QOL) will be assessed with performance status (Karnofsky) and with Lung Cancer Symptom Scale (LCSS) - Observer and patient scale.

CONTACTS AND LOCATIONS:
Overall Officials: Viljem Kovac, MD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia